CLINICAL TRIAL: NCT06494449
Title: A Randomized, Crossover Trial to Assess the Effects of Acute Intake of Meals Containing Higher vs. Lower Energy From Protein on Diet Induced Thermogenesis in Adults With Overweight or Obesity
Brief Title: Effect of Acute Intake of Meals Containing Higher vs. Lower Energy From Protein on DIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2412
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Higher protein (Experimental)
  Interventions: Other: Higher protein
- Lower protein (Active Comparator)
  Interventions: Other: Lower protein

INTERVENTIONS:
Other: Higher protein — An acute mixed meal containing higher protein
  Arms: Higher protein
Other: Lower protein — An acute mixed meal containing lower protein
  Arms: Lower protein

SUMMARY:
The objective of this trial is to assess the effects of acute intake of mixed meals containing higher vs. lower energy from protein on diet induced thermogenesis (DIT) in adults with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 55 years of age, inclusive. There will be approximately equal numbers of men and women within the groups with overweight/obesity and normal weight.
2. Individual has BMI of 18.5 to 24.9 kg/m2 or 27.0 to 34.9 kg/m2, inclusive.
3. Individual has a REE (measured at the screening visit using indirect calorimetry) between 1,250 and 2,250 kcals/d.
4. For premenopausal women, individual has a history of regular menstrual cycles (21-35 d per cycle) for at least 3 months prior to visit 1.
5. Individual is judged by the Investigator to be in generally good health on the basis of medical history and screening measurements.
6. Individual is willing and able to undergo the scheduled study procedures.
7. Individual understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Individual has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
2. Individual has a clinically significant medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results. Health conditions may include history or presence of clinically important cardiac, renal, hepatic, endocrine (i.e., diabetes), pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
3. Use of tobacco/nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1.
4. Use of hemp/marijuana products within 12 months of visit 1. Occasional use (e.g., once or twice a month) within 12 months of visit 1 is allowed but requires at least a 14-d washout prior to visit 1 and the participant must be willing to refrain from use during the study.
5. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.
6. Individual has used an alpha-blocker, beta-blocker, or high-dose diuretic within 30 d of visit 1. Unstable use (initiation or change in dose) within 30 d of visit 1 of other antihypertensive medications is also exclusionary.
7. Unstable use (initiation or change in dose) within 30 d of visit 1 of thyroid hormone replacement medications.
8. Unstable use (initiation or change in dose) within 30 d of visit 1 of sex hormones for contraception.
9. Use of medications or supplements that may influence carbohydrate or fat metabolism, including but not limited to hypoglycemic medications and systemic (intravenous, intramuscular, or oral) or ≥1500 µg/d (topical, inhaled, intranasal, or dermal) corticosteroids within 30 d of visit 1.
10. Use of any weight loss medication within 90 d of visit 1.
11. Use of medications or supplements that may influence heart rate, including but not limited to stimulant medications (e.g., amphetamines, methylphenidates, etc.) within 30 d of visit 1.
12. Individual has a history of cancer in the prior 5 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
13. Individual has had a weight change of ± 4.5 kg (10 lbs) in the previous 3 months.
14. Individual has extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian).
15. Individual is actively following a weight loss diet (even if maintaining body weight).
16. Individual habitually consumes a diet with <10% or ≥ 20% of energy from protein.
17. Individual regularly consumes (≥ 2 times per week) protein supplements (wash out is permitted).
18. Individual has a history of bariatric surgery or is actively attempting to lose or gain body weight.
19. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
20. History of any major trauma or major surgical event within 2 months of visit 1.
21. Individual has signs or symptoms of an active infection of clinical significance or has taken antibiotics within 5 days prior to any visit (washout is permitted for re-scheduling of the clinic visit).
22. Individual has an allergy, sensitivity or intolerance to any components of the study meals.
23. Individual is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
24. Individual has been exposed to any non-registered drug product within 30 days prior to screening.
25. Individual has a current or recent history (within 12 months prior to screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
26. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Diet Induced Thermogenesis (DIT) AUC | Pre-consumption (0 minutes) to 300 minutes
  Change in DIT assessed as the area under the curve (AUC)

SECONDARY OUTCOMES:
DIT niAUC | Pre-consumption (0 minutes) to 300 minutes
  Change in DIT assessed as the net incremental area under the curve (niAUC)
Carbohydrate oxidation | Pre-consumption (0 minutes) to 300 minutes
  Change in carbohydrate oxidation assessed as the AUC and niAUC
Fat oxidation | Pre-consumption (0 minutes) to 300 minutes
  Change in fat oxidation assessed as the AUC and niAUC
Respiratory Exchange Ratio (RER) | Pre-consumption (0 minutes) to 300 minutes
  Change in RER assessed as the AUC and niAUC

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Maki, PhD, Study Director — MB Clinical Research & Consulting, LLC
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No